CLINICAL TRIAL: NCT03224650
Title: Validation of Novel Predictive Score for Patients With Spinal Metastases
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Andrew Schoenfeld, Associate Professor, Brigham and Women's Hospital
Other Study IDs: 2017P000203
Record Dates: First submitted 2017-07-14; First posted 2017-07-21 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Spinal Metastases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Surgical: Patients treated surgically for spinal metastases
- Non-operative: Patients treated non-operatively for spinal metastases
- Expectant: Patients receiving no treatment for spinal metastases

SUMMARY:
The investigators are prospectively validating a prognostic clinical tool that uses a patient's modified Bauer grade, ambulatory status, and pre-operative serum albumin to predict survival, post-treatment morbidity, and functional outcomes in patients with metastatic disease involving the spine.

DETAILED DESCRIPTION:
Recently, the investigators proposed a clinical prediction score that used a patient's modified Bauer grade, ambulatory status, and pre-operative serum albumin as a means to predict long-term survival following spine surgery for metastatic disease. This prognostic utility was developed using one-year mortality as the sole outcome measure. While the scoring system demonstrated many of the necessary attributes of a useful prediction tool, including simplicity, ease of use and clinical utility, it has yet to be validated prospectively and its capacity to predict other peri-operative outcomes, including physical and mental function following intervention, pain relief and the risk of complications, remain incompletely explored. To further evaluate the utility of this prognostic score, the investigators propose a series of three integrated experiments that will prospectively determine its capacity to accurately inform clinical decision making and recommendations for surgery for patients with metastatic spinal disease.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Confirmed diagnosis of cancer with metastatic spread to the mobile spine or sacrum
3. Able to consent for themselves at the time of the intake evaluation
4. Speaks English

   Exclusion Criteria:
5. Primary bone tumors or leukemia
6. Metastases to other visceral or skeletal locations, without involvement of the spine or sacrum
7. History of prior spine surgery for metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spinal metastases
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Survival | Up to 3 years
  Mortality is documented using date of death in medical record
EuroQuol 5-Dimension (EQ5D) profile | Up to 3 years
  Assessment of state of health and physical/mental function
Short-Form (SF)-12 | Up to 3 years
  Assessment of state of health and physical/mental function
Visual Analog Scale (VAS) for pain | Up to 3 years
  Assessment of current level of pain
Patient-Reported Outcomes Measurement Information System (PROMIS) | Up to 3 years
  Assessment of global health

SECONDARY OUTCOMES:
Post-treatment morbidity and readmissions | Up to 3 years
  Post treatment complications and readmissions documented in medical record

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Schoenfeld, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiong GX, Collins JE, Ferrone ML, Schoenfeld AJ. Prospective comparison of one-year survival in patients treated operatively and nonoperatively for spinal metastatic disease: results of the prospective observational study of spinal metastasis treatment (POST). Spine J. 2023 Jan;23(1):14-17. doi: 10.1016/j.spinee.2022.02.004. Epub 2022 Feb 16. No abstract available. PMID 35181541